CLINICAL TRIAL: NCT04367662
Title: Study of the Vascular Compartment and Hypercoagulability During Coronavirus Infection COVID-19
Acronym: COVID'HEMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/0104/OB
Record Dates: First submitted 2020-04-16; First posted 2020-04-29 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: Hemostasis
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with COVID-19 infection (Experimental): Patient with COVID-19 infection hospitalized in a COVID unit
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — blood sampling in hospitalized patient for COVID-19 infection

SUMMARY:
Coronavirus COVID-19 is an emerging virus also called Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Eighty percent of patients are poor or asymptomatic. However, there are major respiratory complications for some patients, requiring intensive care hospitalization and possibly leading to death in 5% of cases. One of the hypotheses put forward is that much of the pathophysiology is due to endothelial dysfunction associated with disseminated intravascular coagulation.

The covid-19 pathology could induce coagulation impairment as observed during sepsis. An increase in D-dimer levels during covid-19 disease is itself associated with excess mortality. While D-dimers are highly sensitive, they are not specific for clotting activity. They may be increased in many other circumstances, particularly in inflammation.

On the other hand, the infection stimulates the release of extracellular vesicles. These vesicles, of multiple cellular origin, are an actor of vascular homeostasis, and participate in the state of hyperactivation of coagulation. They have a major role in the prothrombotic state and the development of coagulopathy associated with sepsis.

The aim of our monocentric prospective study would be to study early and more specific markers of hypercoagulability and markers of routine endothelial dysfunction, as soon as the patient is hospitalized, in order to predict the risk of hospitalization in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient admitted to Rouen University Hospital for documented SARS-Cov-2 infection (PCR Test or CT scan)
* Patient who accept to participate to research after reading the information note
* Patient affiliated with Social Security

Exclusion Criteria:

* Patient under protective guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Clinical worsening (yes/no) of the patient during hospitalization | in the 15 days from admission
D-DIMERS plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Fibrin monomers plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Antithrombin plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Prothrombin Fragment 1 plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Prothrombin Fragment 2 plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Thrombin generation test plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Microvesicles of platelet plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Cross-linked platelets plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Willebrand Factor plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling
Factor VIII plasma levels in blood | 1 hour after admission
  Biological analysis using initial blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Paul BILLOIR, pharmacist, Principal Investigator — University Hospital, Rouen; Véronique LE CAM, MD, Study Director — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No